CLINICAL TRIAL: NCT05946590
Title: The Duration of Exclusive Breastfeeding and Tongue-tie in Neonates.
Brief Title: Breastfeeding Duration and Tongue-tie in Neonates.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Diana Skaaning, Clinical Supervisor, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEC 99694
Record Dates: First submitted 2023-06-29; First posted 2023-07-14 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-04

CONDITIONS: Infant Nutrition Disorders
Keywords: Ankyloglossia; Frenotomy; Infants; Intra-oral vacuum; Breastfeeding
MeSH Terms: conditions — Infant Nutrition Disorders; Ankyloglossia; Breast Feeding | interventions — Oral Frenectomy

STUDY DESIGN:
Intervention Model Description: An exploratory prospective cohort study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Frenotomy (Other): Frenotomy performed by a health care professional
  Interventions: Procedure: Frenotomy

INTERVENTIONS:
Procedure: Frenotomy — Frenotomy in which clipping/incised of the lingual frenulum releases the tongue-tie performed by a health care professional
  Other Names: Frenulum release

SUMMARY:
The goal of this observational study is to examine how performed frenotomy in term-born infants influences the breastfeeding duration. The main questions the study aims to answer are how a suspected tongue-tie, vacuum strength, and breastfeeding may be associated. Families of infants with tongue-tie where frenotomy is suspected will be invited to participate. Intra-oral vacuum measurements before and 5-10 days after frenotomy will be obtained and the breastfeeding status followed for 6 months.

DETAILED DESCRIPTION:
Exclusive breastfeeding is defined as feeding the infant with human breast milk only, except for vitamins, minerals supplements and medicine. It is an official recommendation that infants are exclusively breastfed for 6 months. Approximately 60% and 15% of Danish infants are exclusively breastfed for 4 and 6 months respectively. There are many factors that may interfere with the establishment and duration of breastfeeding.

For the infant, breastfeeding depends on the infant´s ability to seal the oral cavity around the breast and integrate the muscular activities of cheeks, lips, jaw, and tongue. Effectively nutritive sucking occurs due to the application of positive pressure when the tongue moves upwards to express milk, followed by an intra-oral vacuum (vacuum) when the tongue moves downwards and draws milk from the breast by suction. The strength of vacuum affects the effectiveness of milk removal from the breast and regulates the volume of milk. A weak vacuum may, therefore, lead to a shortage of milk transfer, diminished milk supply and early breastfeeding stop. Conversely, was in a recently published study found an association between a high vacuum and infants who were exclusively breastfed for the recommended 6 months.

Difficulties in creating an appropriate vacuum may be related to ankyloglossia, tight frenulum also called tongue-tie, a condition in which the lingual frenulum has anterior attachment near the tip of the tongue and/or are unusually thick, tight, and/or short lingual frenulum. Tongue-tie is often detected when the infant shows signs of difficulties during breastfeeding and/or there is maternal nipple pain. The possible consequence of tongue-tie is insufficient infant weight gain, neonatal dehydration, and shortened breastfeeding duration.

In case of breastfeeding difficulties, it is recommended to evaluate the tongue-tie by the Breastfed Babies Assessment Tool score (TABBY) and depending on this assessment frenotomy may be recommended. The value of both the TABBY score and frenotomy is only poorly validated.

Hypothesis We hypothesise vacuum to increase after frenotomy and, thereby, affect breastfeeding duration positively.

ELIGIBILITY:
Inclusion Criteria:

Infant of an adult mother Delivery after 37 completed gestational weeks. Singleton or twin Infant of a mother who intends to breastfeed. At least one parents speak and write English, Danish, Norwegian, or Swedish.

Exclusion Criteria:

Congenital malformation. Reduced lung function.

Max Age: 49 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Breastfeeding duration | Followed 6 months.
  The duration of exclusive and partial breastfeeding

SECONDARY OUTCOMES:
TABBY score | Before and 5-10 days after performed frenotomy.
  The association between tongue-tie, TABBY score, and vacuum strength.
Delta intra-oral vacuum | Before, within 1 hour after and 5-10 days after performed frenotomy.
  The primary outcome is to investigate any difference in vacuum in infants below 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Diana Skaaning, Principal Investigator — Region Hovedstadens Apotek
Locations (1):
- Diana Skaaning, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
All personal information about potential and enrolled participants will be collected, shared, and maintained under protected confidentiality before, during, and after the study period according to Capital Region at Knowledge Center for Data Reviews and the General Data Protection Regulation.